CLINICAL TRIAL: NCT03325088
Title: Assessing the Expression and the Activity of Rac1 Protein in the Airway Smooth Muscle of
Brief Title: Assessing the Expression and the Activity of Rac1 Protein in the Airway Smooth Muscle of Asthmatic Patient
Acronym: NaRacAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: L'institut du thorax - INSERM UMR 1087 / CNRS UMR6291 - IRS-Université de Nantes (Unknown); IRSR-PL : Institut de Recherche en Santé Respiratoire des Pays de La Loire (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC16_0469
Record Dates: First submitted 2017-10-20; First posted 2017-10-30 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Asthma
Keywords: Severe Asthma; airway smooth muscle cells; Rac1 protein
MeSH Terms: conditions — Asthma | interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Severe Asthma (Other): patients affected with severe asthma s defined by ERS-ATS (European Respiratory Society - American Thoracic Society) without long term oral corticosteroids treatment
  Interventions: Procedure: Bronchial endoscopy; Procedure: Bronchial biopsies; Procedure: Bronchial alveolar enema
- Mild to moderate Asthma (Other): patients affected with untreated mild to moderate asthma
  Interventions: Procedure: Bronchial biopsies; Procedure: Bronchial alveolar enema
- Controlled Sample (Other): smooth muscle cells from Tracheobronchial rings of non-asthmatic cadaveric donor
  Interventions: Procedure: Bronchial biopsies

INTERVENTIONS:
Procedure: Bronchial endoscopy — Bronchial endoscopy will be performed after clinical examination and pulmonary function tests
  Arms: Severe Asthma
Procedure: Bronchial biopsies — 5 biopsies will be done and analysed at the end of recruiting to assess monomeric GTP Rac1 protein expression and activity on bronchial biopsies
Procedure: Bronchial alveolar enema — For participants who had signed ancillary research consent
  Arms: Mild to moderate Asthma; Severe Asthma

SUMMARY:
Asthma is a chronic inflammatory respiratory disease affecting 6 to 7% of the French adult population and responsible of 1000 deaths in France every year. Many anti-inflammatory treatments are available but few had been developed to target hyperresponsiveness.Investigators and searchers of the Institut du thorax have recently demonstrated the main involvement of Rac1 monomeric G protein in the contraction of airway smooth muscle cells. They show that Rac1 is expressed in the airway smooth muscle cells in mice and its activity is increased in the bronchi of asthma induced mice sensitized to House-Dust Mite. They further demonstrate that Rac1 inhibition in mice by nebulisation reduces airway hyperresponsiveness and pulmonary inflammation. Investigators and searchers of the Institut du thorax would like to seek whether targeting Rac1 would be interesting in asthmatic patients. Primary objective of this study is to determine if Rac1 expression and activity in airway smooth muscle cells are increased in asthmatic patients compare to controlled samples (deceased donor samples). Secondary objective is to determine whether there is a correlation between Rac1 activity and asthma severity.

If Rac1 activity in airway smooth muscles is indeed increased in asthmatic patients depending on asthma severity, Rac1 could be a potential target to treat airway hyperresponsiveness.

DETAILED DESCRIPTION:
Patients will be openly labeled in one of the following group

* 15 patients with severe asthma, without oral corticosteroids treatment.,
* 6 patients with mild to moderate asthma without treatment,
* 21 controlled samples from smooth muscle cells of non-asthmatic deceased donor Bronchial endoscopy with bronchial biopsies will be assessed in all asthmatic patients, Control samples will be obtained from tracheobronchial rings of cadaveric donor. Expression and activity of Rac1 in airway smooth muscle will be determined by immuno-staining on paraffinised biopsies.

Patients will undergo two study visits (D0: inclusion visit, D15: exploratory visit) and one phone call at D21.

Inclusion Visit (D0):

* Signature of the Informed consent,
* Medical History,
* Clinical examination,
* Pulmonary Function Test,
* Blood samples for fibroscopy safety,
* ACT (Asthma Control Test), ACQ (Asthma Control Questionnaire), AQLQ (Asthma Quality of Life Questionnaire), Morisky questionnaire

Exploratory visit (D15)

* Clinical examination,
* Bronchial endoscopy with biopsies Adverse event

Phone Call (D21)

- Adverse event

Recruitment will last 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic Patient :

  * Male or Female from 18 to 70 years old,
  * Diagnosis of asthma confirmed by

    * Existence of one or more following symptoms over 3 months at least (wheezing dyspnea, wheezing, chronic cough and tightness in the chest…)
    * AND past pulmonary function test showing a reversible obstructive ventilatory syndrome after inhaled short-acting bronchodilators (improvement of FEV1 above 12% and at least 200 mL FEV1 gain compare to pre-bronchodilatator FEV1)
    * AND a removal of the clinically suspected differential diagnoses of asthma (vocal cord dysfunction, Churg-Strauss syndrome etc…). The comorbidities should have been explored and treated or on treatment at enrollment.
  * Subject agreed to participate to the study and the biological samples collection,
  * Subject is affiliate to a social security system.
* Inclusion criteria for severe asthmatic patient :

Patient with one of the following criterion will be considered as severe asthmatic patient :

* Patient with a controlled asthma but using high dose of inhaled corticosteroids with another therapeutic classes,
* OR Patient with uncontrolled asthma despite treatment,
* OR Patient with worsening asthma despite treatment.

  -->Inclusion criteria for non-severe asthmatic patients :
* Moderate Asthmatic patient without standard of care treatment since at least one week before the exploratory visit.

  -->Controlled sample:
* Non asthmatic cadaveric adults

Exclusion Criteria:

* Asthmatic Patient :

  * Underage,
  * Pregnant or breast-feeding women,
  * Adult on guardianship
  * Active smoker (smoked or Inhaled),
  * former smokers (smoked or Inhaled) with a smoking history of ≥10 pack years since less than 5 years.
  * Patient with asthma exacerbation the 4 past weeks before the exploratory visit..
  * Patient treated by long term oral corticosteroids or ongoing biological therapy or stopped within the 3 months before exploratory visit.
  * Patient with severe acute or chronic organ disorder (cardiovascular, respiratory, hepatic, renal, malabsorption)
  * Patient with history of unstable angina,
  * Patient with platelet count abnormality, or primary or acquired thrombopathy, or an aPTT (activated Partial Thromboplastin Time) greater than or equal to 1,5 times normal or patient with a Quick Time > 26 seconds
  * Patient under a systemic immunomodulatory or immunosuppressive treatment
  * Patient with anticoagulants or anti-platelet aggregating drugs other than D-lysin acetylsalicylate and that could not be suspended before the bronchial fibroscopy.
  * Patient with hypersensitivity to the treatment used during the bronchial fibroscopy: Hydroxyzine, Midazolam, Xylocaine.
  * Patient with AME (Government Medical Assistance),
  * Patient having physical and psychological disabilities to follow the protocol,
  * Patient included in another interventional research protocol,
  * Patient having risk factors of Creutzfeld-Jakob disease
* Controlled sample:

  * Asthmatic patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Activity level and expression of Rac1 protein in airway smooth muscle cells of asthmatics vs non asthmatics samples | at day 15
  Mean of fluorescence intensity of Rac1-GTP and Rac1 in paraffinised biopsies of airway smooth muscle cells

SECONDARY OUTCOMES:
Assessing any difference between activity level and expression of Rac1 in airway smooth muscle cells of severe versus non severe asthmatic patients. | at day 15
  Mean of fluorescence intensity of Rac1-GTP and Rac1 in paraffinised biopsies of airway smooth muscle cells.
Assessing any correlation between Rac1-GTP/Rac1 ratio signal, pulmonary function tests and clinical data | at day 15
  Mean of fluorescence intensity of Rac1-GTP and Rac1 in paraffinised biopsies of airway smooth muscle cells.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No